CLINICAL TRIAL: NCT02461641
Title: The NuTech NuShield and Affinity Membrane Product Evaluation for the Treatment Neuropathic Diabetic Ulcers (DFU)
Brief Title: NuShield/Affinity for the Treatment of Neuropathic Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NuTech Medical, Inc (Industry)
Collaborators: Organogenesis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD2014-08-03
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2018-10

CONDITIONS: Foot Ulcer, Diabetic
Keywords: amniotic tissue; diabetic foot ulcer; Affinity; NuShield
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard of Care (Other): Wounds will be treated with Standard of Care treatment which for the purpose of this study is defined as, extensive debridement of nonviable tissue, saline-moistened non-occlusive dressing and off-loading to decrease press on the extremity using a DARCO shoe.
  Interventions: Other: Standard of Care
- NuShield (Experimental): Wounds will be treated with Standard of Care treatment which for the purpose of this study is defined as, extensive debridement of nonviable tissue, saline-moistened non-occlusive dressing and off-loading to decrease press on the extremity using a DARCO shoe. In addition, wounds will be treated with a dehydrated amnion-chorion membrane, NuShield, for up to 4 weeks.
  Interventions: Other: NuShield
- Affinity (Experimental): Wounds will be treated with Standard of Care treatment which for the purpose of this study is defined as, extensive debridement of nonviable tissue, saline-moistened non-occlusive dressing and off-loading to decrease press on the extremity using a DARCO shoe. In addition, wounds will be treated with a fresh hypothermically stored amniotic membrane, Affinity, for up to 4 weeks.
  Interventions: Other: Affinity

INTERVENTIONS:
Other: NuShield — NuShield is a sterilized dehydrated amnion chorion membrane patch.
  Arms: NuShield
Other: Affinity — Affinity is a aseptically produced hypothermically stored amniotic membrane patch.
  Arms: Affinity
Other: Standard of Care — Standard of Care for this study is defined as sharp debridement, moist wound dressing and offloading of the area using a DARCO shoe.
  Arms: Standard of Care

SUMMARY:
This study was designed to determine the heal rate of diabetic foot ulcers at 4 weeks, and complete closure at 8 and 12 weeks of patients treated with either NuShield or Affinity compared to standard care alone.

DETAILED DESCRIPTION:
This is a three (3)-arm evaluation in 100 patients over 3 facilities with diabetic foot ulcers (DFU). Patients will be treated with NuShield or Affinity together with standard therapy or with standard care alone. For the purposes of this evaluation, standard therapy will consist of extensive debridement of nonviable tissue, saline-moistened non-occlusive dressing, off-loading to decrease pressure on extremity, aggressive treatment of infection and arterial revascularization if indicated. The patients will receive NuShield or Affinity plus standard therapy to determine optimal application method. The evaluation duration is 4 weeks with 8-week and 12-week follow-up visits. Patients with diabetic neuropathic foot ulcers of at least 4 weeks duration and free of clinical signs of infection at the time of treatment may be eligible for inclusion. At Week -1, each patient will undergo aggressive, surgical debridement. The site should be free of fibrin, necrotic and callous tissue. Digital imaging and planimetery of the target ulcer will be performed pre- and post initial debridement and at each subsequent visit as per the evaluation schedule. This evaluation is designed to investigate the potential of an allogeneic placental-derived amniotic membrane to accelerate healing of lower extremity DFU when used in conjunction with standard therapy. This potential will be measured as an increase in the rate of healing (daily decrease in percent wound area/volume compared to initial debrided ulcer area/volume) of patients treated with NuShield or Affinity plus standard wound care compared to patients treated with standard good wound care alone. Studies by Margolis and co-workers have demonstrated that the use of this surrogate marker, measured at 4 and 8 weeks of care, is predictive (>70%) of wound healing in patients with DFU at the 20th week of care. [Kantor 1998; Margolis 2003] The secondary endpoint will be patients achieving complete closure (100%) by week 12.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is or greater than 18 years old.
2. Type 1 or Type 2 diabetes.
3. Subject has plantar ulcers of greater than or equal to 4 weeks duration at presentation, unresponsive to standard wound care.
4. Subject's ulcer size >0.5cm2 and < 20cm2 area post-debridement.
5. Subject has well controlled glucose levels, with HbA1c < 10%.
6. Subject has adequate lower extremity perfusion, with Ankle-Brachial Index > 0.8 (note: this is an ABI-equivalent, based on biphasic or triphasic color duplex - PVR or MRA. Diabetics often have peripheral vascular calcification or poorly compressible vessels resulting in abnormally high Ankle-Brachial Indices.) or dorsum transcutaneous oxygen test (TcPO2) > 30 mmHg. Presence of tibial and plantar pulses is preferred.
7. Subject should have no evidence of unresolved gross soft-tissue infection or boney pathology (i.e. osteomyelitis).
8. Subject should have no evidence of underlying co-morbid conditions that would adversely affect wound healing such as: Cancer, Raynaud's syndrome, severe venous insufficiency or uncorrected arterial insufficiency, etc.
9. Subject should not be on medications that compromise healing: cytotoxic chemotherapeutics, etc

Exclusion Criteria:

1. Patients with evidence of skin cancer within or adjacent to the ulcer site.
2. Patients who have signs and symptoms of boney pathology (i.e. osteomyelitis) following debridement.
3. Patients with ulcers on the calcaneus.
4. Patients who have significant arterial disease as determined by ABI, duplex Doppler sonography (PVR) or magnetic resonance angiography (MRA): Ankle-Brachial Index < 0.8 (note: this is an ABI-equivalent, based on biphasic or triphasic color duplex - PVR or MRA. Diabetics often have peripheral vascular calcification or poorly compressible vessels resulting in abnormally high ABIs); dorsum transcutaneous oxygen test (TcPO2) < 30 mmHg; absence of tibial or plantar pulses.
5. Patients who have documented clinically significant medical conditions, which would impair wound healing. This includes:

   * Renal impairment (creatinine >2.5 mg/dL);
   * Hepatic impairment (2XULN);
   * Hematological disorders (abnormities of formed elements);
   * Neurologic disorders resulting in significant impairment of sensory and motor functions as judged by the investigator;
   * Patients with signs and symptoms of cellulitis;
   * Patients with ulcers with sinus tracts associated with an ongoing infection;
   * Patients with active deep vein thrombosis;
   * Patients with uncontrolled diabetes, as demonstrated by increased HbA1C (> 10%);
   * Immunocompromised patients (e.g., lymphoma, AIDS, myelodysplastic disorders)
   * Patients with a history of basal cell carcinomas or actinically induced squamous cell carcinomas which have been effectively treated are not excluded, except if the skin cancer was in the exact location of the target ulcer.
6. Patients with active systemic cancer receiving active cancer therapy
7. Patients who are currently receiving, or have received within 1 week prior to study entry:

   * Adriamycin (doxorubicin), bleomycin, serolimus (Rapamune, rapamycin) and anti-TNFα cytotoxic/immunosuppressive agents;
   * Radiation therapy at the ulcer site;
   * Topical growth factors at the target site (i.e., Regranex®).
8. Patients enrolled in wound or drug investigational agent study for any disease within the past 4 weeks.
9. Patients previously treated with amniotic membrane, PRP/PRFM, stem cell therapy, Apligraf, OrCel, Dermagraft, Graft Jacket, Oasis, stem cell therapy or any other advanced therapy at the target site for 1 month prior to enrollment.
10. Pregnant or breast-feeding.
11. Patients, who in the opinion of the investigator, for any reason other than those listed above, will not be able to complete the study per protocol.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2015-03; Primary Completion 2018-04-30 (Actual); Study Completion 2018-10-25 (Actual)

PRIMARY OUTCOMES:
Mean adjusted heal rate | 4 weeks
  Percentage change in area method using ARANZ camera

SECONDARY OUTCOMES:
Extent of wound closure at 12 weeks | 12 weeks
  Percentage of wound closed at 12 weeks.
Length of time to 100% healing of foot ulcer | Up to 12 weeks
  Time (in days) to 100% healing-- complete closure in the absence of drainage

CONTACTS AND LOCATIONS:
Overall Officials: Katie Mowry, PhD, Study Director — NuTech Medical, a division of Organogenesis
Locations (7):
- United States (7):
  - Limb Preservation Platform, Fresno, California
  - The Miller Care Group, Indianapolis, Indiana
  - The Wound Treatment Center, Opelousas, Louisiana
  - Wound Institute and Research Center, Dunmore, Pennsylvania
  - Temple University School of Pediatric Medicine, Philadelphia, Pennsylvania
  - Richard C. Galperin, DPM, FAPWCA, Dallas, Texas
  - Futuro clinical Trials, LLC, McAllen, Texas

IPD SHARING:
Plan to Share IPD: No